CLINICAL TRIAL: NCT03941730
Title: Therapeutic Targeting of ER Beta in Triple Negative Breast Cancer
Brief Title: Estradiol in Treating Patients With ER Beta Positive, Triple Negative Locally Advanced or Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1831; P50CA116201 (NIH); R01CA249116 (NIH); NCI-2019-02285 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1831 (Other: Mayo Clinic in Rochester); 18-000734 (Other: Mayo Clinic Institutional Review Board); TBCRC051 (Other: Translational Breast Cancer Research Consortium)
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Advanced Triple-Negative Breast Carcinoma; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Triple-Negative Breast Carcinoma; Recurrent Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — Biopsy; Magnetic Resonance Spectroscopy; Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (estradiol) (Experimental): Patients receive estradiol PO TID for days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo a tissue biopsy at the end of cycle 1, collection of blood samples on C1D1, at the end of cycle 1, and at the end of treatment. In addition, patients undergo CT, MRI, or PET scans at baseline, at the end of cycles 2, 4, and 6, and then every 8 weeks until disease progression.
  Interventions: Procedure: Biopsy; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Biological: Therapeutic Estradiol

INTERVENTIONS:
Procedure: Biopsy — Undergo tissue biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Biological: Therapeutic Estradiol — Given PO
  Other Names: 17 Beta-Estradiol; Aquadiol; Climara; Dimenformon; Diogyn; Diogynets; Estrace; ESTRADIOL; Estraldine; Oestradiol; Ovocylin; Progynon; Vagifem

SUMMARY:
This phase II trial studies how well estradiol works in treating patients with estrogen receptor beta (ER beta) positive, triple negative breast cancer that has spread to nearby tissue or lymph nodes (locally advanced) or other places in the body (metastatic). Hormone receptors like ER beta allow the body to respond appropriately to hormones. Triple negative means that the breast cancer does not express other hormone receptors called ER alpha, progesterone, and HER2. In some people with triple negative breast cancer, ER beta is overexpressed. Tumor cells that overexpress ER beta grow slower in the laboratory and this growth is slowed in the presence of estrogen. Estradiol is a form of estrogen. This study may help doctors determine whether tumor cells that overexpress ER beta shrink in the presence of estradiol.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the anti-tumor activity of estradiol in patients with locally advanced or metastatic triple negative breast cancer (TNBC) that expresses ERbeta (> 25% moderate or strong nuclear staining).

SECONDARY OBJECTIVES:

I. To examine the safety profile of estradiol when administered at a dose of 2 mg three times daily (TID) to women with locally advanced or metastatic TNBC that expresses ERbeta.

II. To examine the changes in phosphorylated (phospho)-ERbeta, cystatins 1, 2, 4 and 5, phospho-Smad2/3 and Ki-67 in tumor biopsies taken before and after the first cycle of treatment.

EXPLORATORY OBJECTIVES:

I. To examine changes in plasma estradiol, serum cytokine and cystatin levels before/after 1 cycle of estradiol.

II. Analyze the global gene expression profiles of paired biopsies prior to and following 1 cycle of therapy.

III. To develop patient derived xenografts (PDX) that are ERalpha negative, HER2 negative and ERbeta positive (Mayo only).

IV. To examine changes in the relative abundance of circulating immune cell populations after the first cycle of treatment and whether these changes differ with respect to whether the patient is still on treatment after 6 cycles of treatment or not.

OUTLINE:

Patients receive estradiol orally (PO) TID for days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo a tissue biopsy at the end of cycle 1, collection of blood samples on day 1 of cycle 1 (C1D1), at the end of cycle 1, and at the end of treatment. In addition, patients undergo computed tomography (CT), magnetic resonance imaging (MRI), or positron emission tomography (PET) scans at baseline, at the end of cycles 2, 4, and 6, and then every 8 weeks until disease progression.

After completion of study treatment, patients are followed up annually for 5 years from study registration.

ELIGIBILITY:
Inclusion Criteria:

* PRE-SCREENING CRITERIA (STEP 0): Women of age >= 18 years
* PRE-SCREENING CRITERIA (STEP 0): History of locally advanced or metastatic breast cancer that is ERalpha negative or low (< 1% nuclear staining) and HER2 negative.

  * Note: HER2 negative disease per 2018 American Society of Clinical Oncology/College of American of Pathologists (ASCO/CAP) guidelines, one of the following must apply:

    * 0 or 1+ by immunohistochemistry (IHC) and not amplified by in situ hybridization (ISH);
    * 0 or 1+ by IHC and ISH not done;
    * 2+ by IHC and ISH results are: < 6.0 HER2 signals/cell with HER2/CEP17 ratio < 2.0;
    * IHC not done and not amplified by ISH.
* PRE-SCREENING CRITERIA (STEP 0): =< 3 prior chemotherapy regimens for treatment of metastatic breast cancer.

  * Note: Prior use of monoclonal antibodies targeting PD1, PDL1 is allowed (if administered as monotherapy it is not counted as a chemotherapy regimen).
* PRE-SCREENING CRITERIA (STEP 0): Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* PRE-SCREENING CRITERIA (STEP 0): Willing to submit a biopsy specimen from locally recurrent or metastatic site (or primary if metastatic site not available) of breast cancer for ERbeta staining to Mayo Clinic Anatomic Pathology.
* PRE-SCREENING CRITERIA (STEP 0): No prior history of metastatic ERalpha positive breast cancer (>= 1%)
* PRE-REGISTRATION CRITERIA (STEP 1): Presence of moderate or strong nuclear ERbeta staining in > 25% of cells in specimen submitted during Pre-Screening Step.
* PRE-REGISTRATION CRITERIA (STEP 1): For patients who did not have a biopsy or lacking ERalpha, progesterone receptor (PR), and HER2 results from a locally advanced or metastatic site performed =< 12 months prior to Pre-Registration: Willing to undergo a standard of care biopsy of locally recurrent or metastatic breast cancer for ERalpha, PR, and HER2 as well as additional research cores.
* PRE-REGISTRATION CRITERIA (STEP 1): Measurable or non-measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria that will be assessed using imaging-based evaluations.

  * Note: The tumor lesion biopsied during the pre-registration period is not considered measurable disease nor a target lesion.
* PRE-REGISTRATION CRITERIA (STEP 1): If history of brain metastases must meet the following criteria:

  * Patients with a history of brain metastases are eligible only if they are asymptomatic and have stable disease for >= 3 months, including < 28 days of prior to pre-registration.
  * Not receiving steroids for brain metastases.
* PRE-REGISTRATION CRITERIA (STEP 1): ECOG performance status 0 or 1.
* PRE-REGISTRATION CRITERIA (STEP 1): =< 3 prior chemotherapy regimens for treatment of metastatic breast cancer.

  * NOTE: Prior use of monoclonal antibodies targeting PD1, PDL1 is allowed.
* PRE-REGISTRATION CRITERIA (STEP 1): Women must be postmenopausal.

  * NOTE: Postmenopausal status is verified by:

    * Prior bilateral surgical oophorectomy, or
    * Age >= 60 years, or
    * Age < 60 years with no menses for > 1 year with estradiol levels within postmenopausal range, according to institutional standard.
* PRE-REGISTRATION CRITERIA (STEP 1): Able to swallow oral medications.
* PRE-REGISTRATION CRITERIA (STEP 1): Willingness to stop use of strong inducers or inhibitors of CYP3A4 prior to registration.

  * NOTE: Use of strong inducers or inhibitors is allowed during pre-registration as long as patient will complete course prior to registration.
* REGISTRATION CRITERIA (STEP 2): For patents who had a biopsy taken from a metastatic site =< 12 months prior to Pre-Registration: Confirmation from the local lab that the tumor from this biopsy was ERalpha negative (< 1% nuclear staining) and HER2 negative
* REGISTRATION CRITERIA (STEP 2): For patients who underwent a pre-registration biopsy: Histologic confirmation from local lab that tumor is ERalpha negative (< 1% nuclear staining), and HER2 negative
* REGISTRATION CRITERIA (STEP 2): Hemoglobin >= 8 g/dL (=< 14 days prior to registration).
* REGISTRATION CRITERIA (STEP 2): Platelet count >= 75,000/mm^3 (=< 14 days prior to registration).
* REGISTRATION CRITERIA (STEP 2): Creatinine =< 1.5 x upper limit of normal (ULN) (=< 14 days prior to registration).
* REGISTRATION CRITERIA (STEP 2): Total bilirubin =< 1.5 x ULN (=< 14 days prior to registration).
* REGISTRATION CRITERIA (STEP 2): Aspartate aminotransferase/serum glutamic-oxaloacetic transaminase (AST/SGOT) =< 2.5 x ULN (=< 14 days prior to registration).

  * For patients with liver metastasis =< 5 x ULN.

Exclusion Criteria:

* PRE-REGISTRATION CRITERIA: Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection.
  * Symptomatic congestive heart failure.
  * Unstable angina pectoris.
  * Uncontrolled symptomatic cardiac arrhythmia.
  * Uncontrolled hypertension (defined as blood pressure > 160/90).
* PRE-REGISTRATION CRITERIA: Deep vein thrombosis / pulmonary embolism (DVT/PE) =< 12 months prior to pre-registration.

  * Note: Patients who are on anticoagulant therapy for maintenance are eligible as long as the DVT and/or PE occurred > 6 months prior to pre-registration, and there is no evidence for active thrombosis (either DVT or PE).
* PRE-REGISTRATION CRITERIA: Stroke =< 6 months prior to pre-registration.
* PRE-REGISTRATION CRITERIA: Two or more episodes of DVT and/or PE =< 5 years prior to pre-registration.
* PRE-REGISTRATION CRITERIA: Abnormal uterine bleeding =< 6 months prior to pre-registration
* PRE-REGISTRATION CRITERIA: History of coagulopathy.
* PRE-REGISTRATION CRITERIA: Other active second malignancy other than non-melanoma skin cancers within 3 years prior to pre-registration.

  * NOTE: A second malignancy is not considered active if all treatment for that malignancy is completed and the patient has been disease-free for >= 3 years prior to pre-registration.
* REGISTRATION CRITERIA: None of the following therapies are allowed =< 14 days prior to registration.

  * Chemotherapy.
  * Immunotherapy.
  * Biologic therapy.
  * Hormonal therapy.
  * Monoclonal antibodies.
  * Anti-HER2 or other "targeted" (e.g. mTOR) therapy.
  * Note: Any adverse events derived from these therapies must be =< grade 2 prior to starting study therapy (exceptions for alopecia).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit rate | 6 months
  A patient is said to have derived clinical benefit rate at the 6 month time point if the patient's disease meets the Response Evaluation Criteria in Solid Tumors (RECIST) for complete response (CR), partial response (PR), or stable disease (SD) for > 6 months following initiation of treatment. The 6 month clinical benefit rate is the percentage of patients who are found to meet the criteria for clinical benefit at least 6 months among all the patients who have started estradiol treatment. As the number of patients with discordant ERbeta findings are expected to be small, a 90% exact binomial confidence interval will be constructed for the proportion of patients who were found to have no to weak ERβbeta expressing metastatic triple-negative breast cancer (TNBC) and who derived clinical benefit rate at the 6 month time point.

SECONDARY OUTCOMES:
Incidence of adverse events | 5 years
  An adverse event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure. All grade 2, 3, 4 or 5 adverse events will be documented and assigned an attribute by treating clinician as to its relationship to treatment. For a given AE, the proportion of patients who report developing a grade 2-5 of this AE are determined. The number of dose reductions per patient and the reasons for the dose reduction are summarized.
Tumor response rate among those patients with measurable disease | 5 years
  The tumor response rate is defined as the 100% time the number of patients with a CR or PR (as defined by the RECIST criteria) on 2 consecutive evaluations at least 8 weeks apart divided by the total number of eligible patients who began study treatment. A 90% binomial confidence interval is constructed for the true response rate.
Progression free survival (PFS) distribution | Up to 5 years
  PFS is defined as the time from registration to the first of the following events: local, regional, or distant recurrence, second primary disease of death due to any cause. The distribution of PFS times will be estimated using the method of Kaplan-Meier.
Overall survival (OS) distribution | Up to 5 years
  OS is defined as the time from registration to death due to any cause. The distribution of survival times are estimated using the method of Kaplan-Meier.
Changes in phospho-ERbeta, cystatins 1, 2, 4 and 5, phospho-Smad2/3 and Ki-67 | 5 years
  Patients undergo tumor biopsies prior to the start of treatment and at completion of cycle 1 treatment. These specimens will be undergoing immunohistochemistry (IHC) staining with the following antibodies: phosphorylated (phospho)-ERbeta, cystatins 1, 2, 4 and 5, phospho-Smad2/3 and Ki-67. For each of these biomarkers, a times series plot are constructed so that an individual patient's data will be represented using the same color for each of the five graphs. These graphs are visually inspected for trends within each of the graphs (variation between individuals) as well as across the five graphs (profile of biomarker changes within an individual).

OTHER OUTCOMES:
Changes in serum cystatin levels in response to treatment | Baseline up to cycle 1
  Change in cystatin levels following one cycle of treatment are examined using signed rank tests and the difference in the percent change in its level following one cycle of treatment between patients who derived clinical benefit and those who did not will be examined using a two sample Wilcoxon rank sum test.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P. Goetz, M.D., Principal Investigator — Mayo Clinic
Locations (9):
- United States (9):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - FHCC South Lake Union, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/30/NCT03941730/ICF_000.pdf